CLINICAL TRIAL: NCT02369419
Title: Frailty Score Assessment for Elderly Patients Undergoing Cardiac Resynchronization Therapy
Acronym: FRAILTY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Rouen (Other); University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2013-02-DR-KUBALA
Record Dates: First submitted 2015-02-16; First posted 2015-02-24 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Heart Failure
Keywords: frailty; Heart failure; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT: Patients over 70 years age, selected for CRT according to the ESC 2013 guidelines.
  Interventions: Other: Frailty

INTERVENTIONS:
Other: Frailty — CRT device is implanted in all patients selected for the study. Frailty is evaluated before implant and defined as <14/17 points using the ONCODAGE score

SUMMARY:
Background: The cardiac resynchronization therapy (CRT) has been shown to improve symptoms and outcome of patients with congestive heart failure (HF), and depressed left ventricular ejection fraction (LVEF < 35 %). The rate of non-responders to CRT is estimated at 30 %. Yet, the impact of frailty on the response to CRT has not been studied, until now.

Purpose : To assess the impact of frailty in the elderly, on the response to CRT.

DETAILED DESCRIPTION:
Methods : Frailty is evaluated before implant ,and defined as <14/17 points using the ONCODAGE score, in 150 patients of > 70 years age, selected for CRT according to the ESC 2013 guidelines. The response to CRT, estimated at 9 months, is defined as an improvement of at least 5 % of the LVEF and the absence of HF hospitalization or cardiovascular death.

ELIGIBILITY:
Inclusion Criteria:

* Patients of > 70 years age,
* Selected for CRT according to the ESC 2013 guidelines

Exclusion Criteria:

* patients included in other clinical trial which can interfere with the results of this one

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of > 70 years age, selected for CRT according to the ESC 2013 guidelines
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
non response on CRT | 9 months

SECONDARY OUTCOMES:
seric albumin | 9 months
  To assess the impact of seric albumin on the response to CRT
seric gammaglutamyltranferase | 9 months
  To assess the impact of seric gammaglutamyltranferase on the response to CRT
mortality | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Maciej KUBALA, Principal Investigator — CHU Amiens
Locations (1):
- CHU; Service de Cardiologie, Rythmologie et Stimulation cardiaque, Amiens, France

REFERENCES:
- [Derived] Kubala M, Guedon-Moreau L, Anselme F, Klug D, Bertaina G, Traulle S, Buiciuc O, Savoure A, Diouf M, Hermida JS. Utility of Frailty Assessment for Elderly Patients Undergoing Cardiac Resynchronization Therapy. JACC Clin Electrophysiol. 2017 Dec 26;3(13):1523-1533. doi: 10.1016/j.jacep.2017.06.012. Epub 2017 Sep 13. PMID 29759834